CLINICAL TRIAL: NCT04217447
Title: Assessment of Quitting Versus Using Aspirin Therapy In Patients Treated With Oral Anticoagulation for Atrial Fibrillation or Other Indication With Stabilized Coronary Artery Disease
Acronym: AQUATIC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The sponsor's decision to stop the study follows the DSMB's recommendations (end of enrolment and experimental treatment, post-treatment/end-of-study visit within 3 months of stopping treatment), regarding the benefit-risk balance.
Sponsor: University Hospital, Brest (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 29BRC19.0116
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease
Keywords: atrial fibrillation; oral anticoagulation; antithrombotic therapy
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: It's a prospective, randomized, double-blind, placebo controlled, parallel-group, multi-center study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Active Comparator): Patients intaking full-dose OAC + ASA 100mg od
  Interventions: Drug: OAC + Aspirin 100mg od
- Control group (Placebo Comparator): Patients intaking full-dose OAC + Placebo of ASA 100mg od
  Interventions: Drug: OAC + placebo of Aspirin 100mg od

INTERVENTIONS:
Drug: OAC + Aspirin 100mg od — Patients will receive full-dose of OAC + Aspirin 100mg od during 24 to 48 months (until death or the end of the study : i.e. achievement of 2-year follow-up of the last included patient, maximum of 48-month followup for the first included patient)
  Arms: Experimental group
Drug: OAC + placebo of Aspirin 100mg od — Patients will receive full-dose of OAC + placebo of Aspirin 100mg od during 24 to 48 months (until death or the end of the study : i.e. achievement of 2-year follow-up of the last included patient, maximum of 48-month followup for the first included patient)
  Arms: Control group

SUMMARY:
* Long-term aspirin (ASA) is the standard recommended antithrombotic therapy in patients with stable coronary artery disease (CAD), especially following stenting (Class I, Level A).
* Long-term oral anticoagulation (OAC) is the standard antithrombotic therapy in patients with atrial fibrillation (AF) associated with one or more risk factor for stroke (Class I, Level A).
* During the first year following acute coronary syndrome (ACS) and/or percutaneous coronary intervention (PCI), several studies evaluating the combination of OAC treatment and antiplatelet therapy are either already published or ongoing.
* At distance of the index ACS and/or PCI, patients with stable CAD and concomitant AF remain at particular high-risk of ischemic (3 to 4 times higher as compared to patients with stable CAD without AF) and bleeding events. Antithrombotic management of these patients is subsequently highly challenging in clinical practice. The European task force suggests that the use of a full-dose anticoagulant monotherapy without any antiplatelet therapy should be the default strategy in such patients with both, AF and stable CAD.
* However, evidences are sparse and weak to support such a strategy (only observational studies with many biases) and no randomized trial has assessed this question. These patients, especially those at high-risk of recurrent ischemic events (post- ACS, diabetes, multivessel CAD…) may benefit from the combination of OAC and aspirin at long-term. Indeed the crude event rate of ischemic events is much higher than the crude event rate of bleeding in this specific population. Ischemic events are 2 to 3 times more frequent than bleeding in daily practice.
* The benefit/risk ratio of these two different strategies (ASA in combination with OAC vs. OAC alone) in patients at high-risk of recurrent coronary and vascular events remains unknown. Dual therapy with full-dose anticoagulation and ASA may lead to higher risk of major bleeding, while stopping ASA in stabilized high-risk patients after PCI may lead to poorer outcome regarding ischemic events.
* The coordinating investigators therefore designed a double blind placebo controlled trial in order to assess the optimal antithrombotic regimen that should be pursued long-life in this subset of patients.

DETAILED DESCRIPTION:
* Long-term aspirin (ASA) is the standard recommended antithrombotic therapy in patients with stable coronary artery disease (CAD), especially following stenting (Class I, Level A).
* Long-term oral anticoagulation (OAC) is the standard antithrombotic therapy in patients with atrial fibrillation (AF) associated with one or more risk factor for stroke (Class I, Level A).
* During the first year following acute coronary syndrome (ACS) and/or percutaneous coronary intervention (PCI), several studies evaluating the combination of OAC treatment and antiplatelet therapy are either already published or ongoing.
* At distance of the index ACS and/or PCI, patients with stable CAD and concomitant AF remain at particular high-risk of ischemic (3 to 4 times higher as compared to patients with stable CAD without AF) and bleeding events. Antithrombotic management of these patients is subsequently highly challenging in clinical practice. The European task force suggests that the use of a full-dose anticoagulant monotherapy without any antiplatelet therapy should be the default strategy in such patients with both, AF and stable CAD.
* However, evidences are sparse and weak to support such a strategy (only observational studies with many biases) and no randomized trial has assessed this question. These patients, especially those at high-risk of recurrent ischemic events (post- ACS, diabetes, multivessel CAD…) may benefit from the combination of OAC and aspirin at long-term. Indeed the crude event rate of ischemic events is much higher than the crude event rate of bleeding in this specific population. Ischemic events are 2 to 3 times more frequent than bleeding in daily practice.
* The benefit/risk ratio of these two different strategies (ASA in combination with OAC vs. OAC alone) in patients at high-risk of recurrent coronary and vascular events remains unknown. Dual therapy with full-dose anticoagulation and ASA may lead to higher risk of major bleeding, while stopping ASA in stabilized high-risk patients after PCI may lead to poorer outcome regarding ischemic events.

AQUATIC is a prospective, randomized, double-blind, placebo controlled, parallel-group, multi-center study.

Randomization into 2 treatment groups and stratified on study center, type of OAC (VKA vs. DOAC), antithrombotic treatment received at the time of inclusion (dual therapy combining single antiplatelet therapy + OAC vs. OAC alone).

Experimental group : Patients intaking full-dose OAC + ASA 100mg od.

Control group : Patients intaking full-dose OAC + Placebo of ASA 100mg od.

Note:

* For Apixaban: in case of > 1 of the followings: > 80 years old, weight < 60kg, creatinine level > 133μmol/l; Or a creatinine clearance between 30 and 50 ml/min (Cockroft Formula), the dose of Apixaban will be reduced to 2.5 mg bid.
* For Rivaroxaban: in case of moderate creatinine clearance (Cockroft Formula) (between 30 and 50 ml/min) or severe renal insufficiency (between 15 and 29 ml/min) the dose of Rivaroxaban will be reduced to 15 mg od.
* For Dabigatran: in case of moderate creatinine clearance (Cockroft Formula) (between 30 and 50 ml/min) with age between 75 and 80 years: the dose of Dabigatran will be 150 mg bid or 110 mg bid, according to the ischemic and hemorrhagic risk of the patient. In case of age > 80 years and/or concomitant administration of Verapamil, the dose of Dabigatran will be reduced to 110 mg bid.
* For VKA: target INR (International Normalised Ratio) between 2 and 3.

The primary efficacy objective is to demonstrate, in high-risk stabilized patients after PCI requiring also anticoagulation for AF, the superiority of the dual therapy ASA 100mg od + full-dose of OAC for 24-48 months versus full-dose of OAC alone (+ placebo) on a composite endpoint associating: cardio-vascular (CV) mortality, myocardial infarction, stroke, coronary revascularization, systemic embolism, and acute limb ischemia.

The primary safety objective is major bleeding (ISTH : International Society of Thrombosis and Haemostasis).

The secondary efficacy objectives are evaluation of efficacy of dual therapy SA 100mg od + OAC full ose versus OAC alone (+placebo) for:

* The composite of CV mortality, MI (Myocardial Infarction ), stroke
* CV mortality
* All cause death
* Myocardial infarction (MI)
* Stent thrombosis (definite or probable)
* Stroke (ischemic, hemorrhagic, or stroke of uncertain cause, transient ischemic attack [TIA])
* Coronary revascularization
* Systemic embolism
* Acute limb ischemia

Net clinical benefit:

* All cause mortality
* Major bleeding [define according to the International Society of Thrombosis and Haemostasis (ISTH): an acute, linically overt bleeding accompanied by one or more of the following findings: 2g/dl decline in Hemoglobin level r = 2 red blood cell transfusions over a 24-hour period, leeding of a major organ (intracranial, intramedullary, intraocular, pericardial, interarticular, intramuscular and / or retro peritoneal) or fatal bleeding]
* Thrombotic cardiovascular events:

  * Myocardial infarction
  * Stent thrombosis
  * Stroke (ischemic, hemorrhagic, or stroke of uncertain cause, TIA)
  * Any coronary revascularization
  * Systemic embolism
  * Acute limb ischemia

The secondary safety objectives are :

* Major and clinically relevant non major bleeding (ISTH)
* Major bleeding (TIMI : Thrombolysis In Myocardial Infarction)
* Major bleeding (BARC ≥3 : Bleeding Academic Research Consortium)

All the included patients will be randomized at visit 1 and followed every 6 months until death or the end of the study (i.e. achievement of 2-year follow-up of the last included patient, maximum of 48 month followup for the first included patient).The first patient may require up to 9 visits .

2000 patients are expected to be included.

Inclusion period : 72 months. Duration of patient's participation: 24 to 48 months depending of time of inclusion.

Total study duration: 48 months.

All included patients will remain in the study until death or the end of the trial (i.e. achievement of 2-year follow-up of the last included patient).

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 year-old
* All patients that need anticoagulation with direct oral anticoagulant (DOAC) or vitamin K antagonist (VKA) for AF (paroxysmal, persistent or permanent) or other indication and have a stabilized CAD (free from MI, or coronary revascularization in the past year) but remain at high residual risk of recurrent coronary and vascular events. The use of DOAC will be promoted as recommended by guidelines.
* Two different categories of patients could be included in the study, i) patients treated at the time of inclusion with the association of OAC and single antiplatelet therapy, it will be tested for them aspirin vs. interruption of antiplatelet therapy ii) patients treated with OAC alone at the time of inclusion, it will be tested for them administration of aspirin vs. no additional treatment with aspirin.
* High-risk of coronary and vascular event is defined as follow :

  1. History of PCI during an ACS involving placement of ≥1 stent(s) since >6 months.
  2. History of PCI (>6 months) outside the context of ACS but with high-risk features of ischemic event recurrences defined as: diabetes, or diffuse multivessel disease (defined by the involvement of the 3 coronary vessels), or chronic kidney disease (creatinine clearance < 50ml/min), or prior stent thrombosis, or complex PCI (defined by: stenting of the last remaining patent coronary artery, left main, at least 3 stents implanted and/or 3 lesions treated, bifurcation with two stents, length of stent >60mm and chronic total coronary occlusion) or the presence of peripheral artery disease (previous limb revascularization bypass or percutaneous angioplasty, previous limb or foot amputation for arterial vascular disease, history of intermittent claudication of peripheral artery stenosis (≥50%) ,previous carotid revascularization or carotid stenosis ≥50%).
* Women of childbearing potential with effective contraception defined as

  * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation :

    * oral
    * intravaginal
    * transdermal
  * progestogen-only hormonal contraception associated with inhibition of ovulation :

    * oral
    * injectable
    * implantable
  * intrauterine device (IUD)
  * intrauterine hormone-releasing system ( IUS)
  * bilateral tubal occlusion
  * vasectomised partner
  * sexual abstinence

Exclusion Criteria:

* Any coronary event within 6 months prior to randomization
* High risk of bleeding defined as recent (≤6 months) ISTH major bleeding event
* Constitutional or acquired haemorrhagic disease including gastrointestinal bleeding and thrombocytopenia
* Planned PCI within the next 6 months after randomization or subject requiring P2Y12 receptor antagonist therapy
* Stroke within 1 month or any history of hemorrhagic stroke
* Any contraindication to aspirin (ASA) or any of these excipients or other NSAIDs (hypersensitivity, allergy, active bleeding)
* Any contraindication to anticoagulant
* History (s) of asthma induced by the administration of salicylates or substances of close activity (especially NSAIDs)
* Evolutionary gastroduodenal ulcer
* Any other gastroduodenal history
* Severe renal insufficiency
* Severe hepatic insufficiency
* Severe, uncontrolled heart failure
* Lactose intolerance
* Pregnancy
* Breastfeeding patients
* Unable (protected adults : tutorship, curatorship) orunwilling to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 874 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Primary efficacy outcome : rate of composite of cardiovascular mortality and thrombotic cardiovascular events | within 24-48 months
  The primary efficacy outcome is the incidence of the adjudicated composite of (within 24-48 months):
  * CV mortality
  * Thrombotic cardiovascular events
    * Myocardial infarction
    * Stroke
    * Any coronary revascularization
    * Systemic embolism
    * Acute limb ischemia
  An Independent Clinical Events Committee (ICEC) will adjudicate all events (ischemic and bleeding events).
Primary safety outcome : rate of major bleeding | within 24-48 months
  The primary safety outcome is the occurrence of major bleeding according to the ISTH (International Society of Thrombosis and Haemostasis) definition

SECONDARY OUTCOMES:
Secondary efficacy outcomes : rate of composite of CV mortality, MI, stroke; CV mortality; all cause of death; thrombotic cardiovascular events. | within 24-48 months
  The secondary efficacy outcomes are the occurrence of any of the following events:
  * The composite of CV mortality, MI, stroke
  * CV mortality
  * All cause death
  * Thrombotic cardiovascular events:
    * Myocardial infarction
    * Stent thrombosis alone (definite or probable)
    * Stroke (ischemic, hemorrhagic, or stroke of uncertain cause, TIA)
    * Any coronary revascularization
    * Systemic embolism
    * Acute limb ischemia
Secondary safety outcomes : rate of major and clinically relevant non major bleeding | within 24-48 months
  The secondary safety outcome are the occurrence of :
  Major and clinically relevant non major bleeding according to the ISTH definition (ISTH : International Society of Thrombosis and Haemostasis) Major bleeding (TIMI : Thrombolysis in Myocardial Infarction) Major bleeding (BARC ≥3 : Bleeding Academic Research Consensus)

CONTACTS AND LOCATIONS:
Locations (51):
- France (51):
  - CHRU d'Amiens, Amiens, France
  - CHU d'Angers, Angers, France
  - CH d'Annecy-Genevois, Annecy, France
  - CH d'Antibes, Antibes, France
  - CH d'Arras, Arras, France
  - CH d'Avignon, Avignon, France
  - CH de la Côte Basque - Bayonne, Bayonne, France
  - Hôpital Haut Lévêque -CHU Bordeaux-Pessac, Bordeaux, France
  - CHU de Brest, Brest, France
  - Hôpital Louis Pradel - Bron, Bron, France
  - Centre Hospitalier René Dubos - Cergy Pontoise, Cergy-Pontoise, France
  - CH Chalon sur Saône, Chalon-sur-Saône, France
  - CH Louis Pasteur - Chartres - Le Coudray, Chartres, France
  - CHU de Clermont-Ferrand, Clermont-Ferrand, France
  - CH Compiègne, Compiègne, France
  - CH Sud Francilien Corbeil-Essonnes, Corbeil-Essonnes, France
  - Hôpital Henri Mondor - Créteil, Créteil, France
  - CHU de Dijon, Dijon, France
  - GHM - Grenoble, Grenoble, France
  - CHU de Grenoble, Grenoble, France
  - Clinique St Clothilde -La Réunion, La Réunion, France
  - CH de Lens, Lens, France
  - CHRU de Lille, Lille, France
  - CHU de Limoges, Limoges, France
  - CH St Joseph-St Luc Lyon, Lyon, France
  - Marseille-Hôpital Nord, Marseille, France
  - Marseille- Hôpital La Timone, Marseille, France
  - CH Martigues, Martigues, France
  - CHU de Montpellier, Montpellier, France
  - Clinique du Millénaire - Montpellier, Montpellier, France
  - CHU de Nîmes, Nîmes, France
  - CHR d'Orléans, Orléans, France
  - Paris-Lariboisière, Paris, France
  - Paris-Pitié-Salpêtrière, Paris, France
  - Paris-HEGP Cardiologie, Paris, France
  - Paris-HEGP Médecine vasculaire, Paris, France
  - Paris-Bichat, Paris, France
  - CH de Pau, Pau, France
  - CH Périgueux, Périgueux, France
  - CHU de Poitiers, Poitiers, France
  - CHU de Rennes, Rennes, France
  - Clinique St Hilaire - Rouen, Rouen, France
  - CHU de Rouen, Rouen, France
  - CH de Seclin, Seclin, France
  - Clinique Rhena - Strasbourg, Strasbourg, France
  - CHU de Strasbourg, Strasbourg, France
  - CHU de Toulouse, Toulouse, France
  - Clinique Pasteur-Toulouse, Toulouse, France
  - CHRU de Tours, Tours, France
  - Hôpital André Mignot - CH de Versailles, Versailles, France
  - CHU de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemesle G, Didier R, Steg PG, Simon T, Montalescot G, Danchin N, Bauters C, Blanchard D, Bouleti C, Angoulvant D, Andrieu S, Vanzetto G, Kerneis M, Decalf V, Puymirat E, Mottier D, Diallo A, Vicaut E, Gilard M, Cayla G; AQUATIC Trial Investigators. Aspirin in Patients with Chronic Coronary Syndrome Receiving Oral Anticoagulation. N Engl J Med. 2025 Oct 23;393(16):1578-1588. doi: 10.1056/NEJMoa2507532. Epub 2025 Aug 31. PMID 40888725